CLINICAL TRIAL: NCT01316224
Title: Prevalence and Incidence of Articular Symptoms and Signs Related to Psoriatic Arthritis in Patients With Psoriasis Severe or Moderate With Adalimumab Treatment
Acronym: TOGETHER
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-598
Record Dates: First submitted 2011-02-14; First posted 2011-03-16 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: Psoriasis; Incidence; Quality of Life; Psoriatic Arthritis; Prevalence
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate or severe plaque psoriasis: Participants with moderate or severe plaque psoriasis treated with adalimumab

SUMMARY:
Psoriatic Arthritis (PsA) is a comorbidity that affects a significant proportion of participants with moderate or severe psoriasis. The purpose of this study was to describe the profile of patients with moderate or severe plaque psoriasis (Ps) in Colombia and to evaluate adalimumab efficacy and safety profile.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disease affecting 1% to 3% of the population worldwide. A significant portion (5%-40%) of participants with psoriasis develop PsA, a chronic inflammatory arthritis that causes progressive joint damage, reduced functionality and increased mortality risk. Skin disease typically manifests before arthritis in more than 80% of PsA participants, and psoriasis symptoms usually precede joint symptoms by an average of 10 years. Participants with psoriasis who have comorbid PsA incur substantially increased cost of care and experience greater impairment of physical functioning and quality of life compared with participants with psoriasis alone.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a documented clinical diagnosis of psoriasis, as determined by participant interview of his/her medical history and confirmation of diagnosis through physical examination by the investigator
* Participant has indication of psoriasis systemic therapy
* If female, participant is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:
* Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
* Contraceptives (oral or parenteral) for three months (90 days) prior to study drug administration
* A vasectomized partner
* Total abstinence from sexual intercourse
* Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* Participants who have active infections
* Participants enrolled in another study or clinical trial
* Any condition that according to the criteria of the participating investigator represents an obstacle for study conduction and/or participants to an unacceptable risk
* History of active tuberculosis (TB), histoplasmosis or listeriosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants treated with adalimumab, per approved label, with moderate or severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel G Uribe, Study Director — Abbvie SAS
Locations (15):
- Colombia (15):
  - Site Reference ID/Investigator# 48347, Barranquilla
  - Site Reference ID/Investigator# 48349, Barranquilla
  - Site Reference ID/Investigator# 53045, Barranquilla
  - Site Reference ID/Investigator# 53047, Bogotá
  - Site Reference ID/Investigator# 78533, Bogotá
  - Site Reference ID/Investigator# 48345, Cali
  - Site Reference ID/Investigator# 48346, Cali
  - Site Reference ID/Investigator# 59342, Cali
  - Site Reference ID/Investigator# 48342, Cartagena
  - Site Reference ID/Investigator# 48348, Cartagena
  - Site Reference ID/Investigator# 53050, Cartagena
  - Site Reference ID/Investigator# 48351, Medellín
  - Site Reference ID/Investigator# 48353, Medellín
  - Site Reference ID/Investigator# 53046, Medellín
  - Site Reference ID/Investigator# 53049, Medellín

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate or Severe Psoriasis: Participants with moderate or severe psoriasis in treatment with adalimumab
Period: Overall Study
Arm/Group | Moderate or Severe Psoriasis
Started | 52
Completed Visit 1 to Dermatologist | 52
Completed Visit 1 to Rheumatologist | 49
Completed Visit 2 to Dermatologist | 51
Completed Visit 3 to Dermatologist | 48
Completed Visit 3 to Rheumatologist | 39
Completed Visit 4 to Dermatologist | 42
Completed Visit 4 to Rheumatologist | 28
Completed | 42
Not Completed | 10
Not completed — Protocol Violation | 3
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event With Treatment Failure | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.85 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants who indicated more than one race are referred to as "Metis"
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 18
    More than one race | 34
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Colombia | 52
Weight [Mean (Standard Deviation); unit: kg] | 78.70 (14.70)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (5.06)
C-Reactive Protein (CRP) (N=10) [Mean (Standard Deviation); unit: mg/dl] — Data is based on available information.
  mg/dl | 1.39 (1.63)
Study Specific Characteristic [Number; unit: Participants] — Participants with family history of PsA is based on available information from participants who completed the visits to the rheumatologist.
  Participants
    Participants Who Smoke | 21
    Positive History of Comorbidities | 28
    Presence of Metabolic Syndrome | 8
    Presence of Hypertension | 15
    Presence of Family History of PsA (N=49) | 11
    Prior Methotrexate Use | 36
    Current Methotrexate Use | 11
    Prior Biologic Therapy | 14

OUTCOME MEASURES:

1. Secondary Outcome: Mean Time to First Occurrence of PsA Signs or Symptoms
Description: The measure of time from Psoriasis diagnosis to the appearance of PsA signs or symptoms.
Time Frame: Baseline up to Visit 4 (month 12)
Population: Participants who completed at least one of the follow up visits to the rheumatologist.
Measure: Mean (95% Confidence Interval); unit: Years
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 44
Years | 23.17 [16.33 to 30.01]

2. Secondary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: The PASI score was used to measure the severity of psoriasis. It combined the assessment of the severity of lesions and the area affected into a single score ranging from 0 (no disease) to 72 (maximal disease).
Time Frame: At Baseline, Visit 2 (month 2), Visit 3 (month 6) and Visit 4 (month 12)
Population: ITT population
Measure: Mean (Standard Deviation); unit: PASI score
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 52
PASI score
  Baseline | 17.42 (12.11)
  Change from Baseline at Visit 2 (N=51) | -11.56 (11.96)
  Change from Baseline at Visit 3 (N=47) | -13.12 (12.69)
  Change from Baseline at Visit 4 (N=41) | -15.17 (12.69)

3. Secondary Outcome: Percentage of Participants With Comorbidities Who Did or Did Not Develop PsA
Description: Percentage of participants with comorbidities (metabolic syndrome, hypertension, diabetes, atherosclerosis, obesity, alcohol and other associated comorbidities) was assessed.
Time Frame: Baseline up to Visit 4 (month 12)
Population: Participants who completed at least one of the follow up visits to the rheumatologist.
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 44
Percentage of participants
  Non-PsA participants (N=25) | 60.0
  PsA participants (N=19) | 52.6

4. Secondary Outcome: Mean Change in Quality of Life (QoL)
Description: The Short Form-36 was a self-reported questionnaire used to measure the QoL of participants in eight main health dimensions (physical functioning; bodily pain; role limitations due to physical health, personal, and emotional problems; emotional well-being; social functioning; vitality; and general health perception). The score from each health dimension was added together for a QoL score on a scale of 0 - 100; a higher score indicated a better QoL.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 52
Score on scale
  Physical Functioning (PF) at Baseline | 78.46 (28.66)
  Change from Baseline in PF at Visit 3 (N=47) | -1.52 (25.80)
  Change from Baseline in PF at Visit 4 (N=47) | -0.95 (24.92)
  Role-Physical (RP) at Baseline | 68.75 (26.89)
  Change from Baseline in RP at Visit 3 (N=47) | 6.52 (26.67)
  Change from Baseline in RP at Visit 4 (N=42) | 6.55 (35.16)
  Bodily Pain (BP) at Baseline (N=51) | 66.78 (29.73)
  Change from Baseline in BP at Visit 3 (N=47) | -0.87 (32.08)
  Change from Baseline in BP at Visit 4 (N=42) | 9.10 (34.82)
  General Health (GH) at Baseline | 57.88 (23.55)
  Change from Baseline in GH at Visit 3 (N=46) | 8.24 (28.30)
  Change from Baseline in GH at Visit 4 (N=42) | 12.95 (31.45)
  Vitality at Baseline | 60.58 (24.37)
  Change from Baseline in vitality at Visit 3 (N=47) | 2.13 (24.18)
  Change from Baseline vitality at Visit 4 (N=42) | 5.51 (30.78)
  Social Functioning (SF) at Baseline | 66.35 (31.07)
  Change from Baseline in SF at Visit 3 (N=47) | 13.56 (29.24)
  Change from Baseline in SF at Visit 4 (N=42) | 13.39 (36.98)
  Role-Emotional (RE) at Baseline | 68.11 (28.47)
  Change from Baseline in RE at Visit 3 (N=47) | 6.03 (29.47)
  Change from Baseline in RE at Visit 4 (N=42) | 15.67 (34.05)
  Mental Health (MH) at Baseline | 64.13 (25.70)
  Change from Baseline in MH at Visit 3 (N=47) | 6.28 (24.33)
  Change from Baseline in MH at Visit 4 (N=42) | 5.45 (30.73)

5. Secondary Outcome: Mean Change in ClASsification Criteria for Psoriatic ARthritis (CASPAR) Score
Description: The CASPAR criteria permits the diagnosis of PsA in spite of low rheumatoid factor positivity. To be classified as having PsA, a participant must have inflammatory articular disease (joint, spine, entheseal) with greater than or equal to 3 of the following 5 points: evidence of psoriasis (current, history of, or family history of); psoriatic nail dystrophy; a negative RF test result; dactylitis (history of or current); and radiographic evidence of juxa-articular new bone formation. Only current psoriasis (2 points) was weighted more heavily than the other features (1 point). CASPER scores range from 1 to 6, with 6 indicating a more definitive diagnosis of PsA.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: Participants who completed the visits (visit 3 and visit 4) to the rheumatologist and for whom information was available.
Measure: Mean (Standard Deviation); unit: CASPAR score
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
CASPAR score
  Baseline | 2.82 (0.73)
  Change from Baseline at Visit 3 (N=38) | 0.05 (0.73)
  Change from Baseline at Visit 4 (N=27) | -0.07 (0.83)

6. Secondary Outcome: Percentage of Participants With a CASPAR Score Greater Than or Equal to 3 at Each Visit to the Rheumatologist
Description: The CASPAR criteria permits the diagnosis of PsA in spite of low rheumatoid factor positivity. To be classified as having PsA, a participant must have inflammatory articular disease (joint, spine, entheseal) with greater than or equal to 3 of the following 5 points: evidence of psoriasis (current, history of, or family history of); psoriatic nail dystrophy; a negative RF test result; dactylitis (history of or current); and radiographic evidence of juxa-articular new bone formation. Only current psoriasis (2 points) was weighted more heavily than the other features (1 point).
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
Percentage of participants
  Baseline | 67.30
  Visit 3 (N=39) | 64.10
  Visit 4 (N=28) | 71.40

7. Secondary Outcome: Percentage of Participants With Swollen Joint Count (SJC) and Tender Joint Count (TJC) Greater Than Zero
Description: Pressure and joint manipulation by physical examination on 68 or 66 joints or regions (34 or 32 per body side, hip joints excluded) were assessed for TJC or SJC, respectively. Both joint tenderness and swelling were classified as present ("1"), absent ("0"), replaced ("9"), or no assessment ("NA"). The total TJC or SJC was derived as the sum of the tender and swollen joints; the range for TJC and SJC was 0 - 68 and 0 - 66, respectively; with higher scores indicating worse conditions.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
Percentage of participants
  SJC at Baseline | 24.50
  SJC at Visit 3 (N=39) | 12.80
  SJC at Visit 4 (N=28) | 7.10
  TJC at Baseline | 36.70
  TJC at Visit 3 (N=39) | 20.50
  TJC at Visit 4 (N=28) | 14.30

8. Secondary Outcome: Percentage of Participants With Joint Symptoms
Description: Joint symptoms were evaluated by presence or absence of peripheral arthritis, morning stiffness and participant reported joint symptoms.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
Percentage of participants
  Baseline | 61.20
  Visit 3 (N=39) | 30.80
  Visit 4 (N=28) | 25.00

9. Primary Outcome: Percentage of Participants Who Developed Psoriatic Arthritis (PsA)
Description: A participant is said to have PsA if they meet the following criteria:
  1. PsA defined by a rheumatologist; or
  2. A participant with inflamed joints >0 and CASPAR score >=3; or
  3. Participant meeting at least one of the two previous definitions.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
Percentage of participants
  Definition 1 - Visit 3 (N=38) | 47.4
  Definition 1 - Visit 4 (N=28) | 35.7
  Definition 2 - Baseline | 17.3
  Definition 2 - Visit 3 (N=39) | 10.3
  Definition 2 - Visit 4 (N=28) | 3.6
  Definition 3 - Visit 3 (N=39) | 46.2
  Definition 3 - Visit 4 (N=28) | 35.7

10. Primary Outcome: Percentage of Participants Who Developed Signs or Symptoms of PsA
Description: Signs or symptoms were defined as mentioning at the rheumatologist visit any joint symptoms prior to or during the visit or a total number of inflamed joints greater than 0.
Time Frame: At Baseline, Visit 3 (month 6) and Visit 4 (month 12)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 49
Percentage of participants
  Baseline | 61.2
  Visit 3 (N=39) | 33.3
  Visit 4 (N=28) | 25.0

11. Secondary Outcome: Incidence Rate of PsA Since Psoriasis Diagnosis
Description: The number of new PsA cases were determined by:
  1. PsA defined by a rheumatologist; or
  2. A participant with inflamed joints >0 and CASPAR score >=3; or
  3. Participant meeting at least one of the two previous definitions occurring over person time (defined as the overall sum of Psoriasis disease duration without PsA).
Time Frame: Baseline up to Visit 4 (month 12)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: new PsA cases per 100 person years
Arm/Group | Moderate or Severe Psoriasis
Number analyzed (Participants) | 52
new PsA cases per 100 person years | 2.66 [1.70 to 4.14]

12. Secondary Outcome: Change in the Subject Proportion That Achieved a PASI (Psoriasis Area and Severity Index) Reduction of ≥50%
Description: This outcome measure was not calculated.
Time Frame: At Baseline, Week 24, and Week 48
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing of informed consent until 70 days or 5 half-lives of drug
Arm/Group | Moderate or Severe Psoriasis
Serious Adverse Events (participants affected / at risk) | 16/52
Other Adverse Events (participants affected / at risk) | 5/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate or Severe Psoriasis (N=52)
Anemia (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
General physical health deterioration (General disorders) | 1
Localised oedema (General disorders) | 1
No therapeutic response (General disorders) | 1
Pain (General disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Tonsillitis bacterial (Infections and infestations) | 1
Alpha 1 fetoprotein increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Breast calcifications (Reproductive system and breast disorders) | 1
Mammary duct ectasia (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 2
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash generalized (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Mastectomy (Surgical and medical procedures) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate or Severe Psoriasis (N=52)
Influenza like illness (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.